CLINICAL TRIAL: NCT04429282
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Intravenous Ibuprofen 400 and 800 mg Every 6 Hours in the Management of Postoperative Pain.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yi Feng, MD (Other)
Responsible Party: Sponsor-Investigator, Yi Feng, MD, Director of department of anesthesiology and painmanagement, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017PHA019
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Ibuprofen; Nonsteroidal Anti-inflammatory Drug; Intravenous; Injectable; Pain; Analgesic
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ibuprofen( 400mg group) (Experimental): Patients were randomly divided into the group received respectively IV ibuprofen 400 mg .
  Interventions: Drug: ibuprofen
- ibuprofen( 800mg group) (Experimental): Patients were randomly divided into the group received respectively IV ibuprofen 800 mg.
  Interventions: Drug: ibuprofen
- placebo group (Placebo Comparator): Patients were randomly divided into the group received respectively IV placebo,.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibuprofen — Patients were randomly divided into three groups in radio 1:1:1 received respectively IV placebo, ibuprofen 400 mg or ibuprofen 800 mg. The first dose of study drugs was administered intravenously at the time of wound closure and then every 6 hours within 48 hours after the operation.
  Arms: ibuprofen( 400mg group); ibuprofen( 800mg group)
Drug: Placebo — Placebo
  Arms: placebo group

SUMMARY:
This study was to evaluate the efficacy and safety of intravenously administered ibuprofen 400mg and 800 mg q6h for the management of moderate to severe postoperative pain in Chinese population.

DETAILED DESCRIPTION:
This randomized, parallel, double-blind, placebo controlled multi-center clinical study was conducted in 396 patients scheduled to undergo elective general anesthesia laparotomy or orthopedic surgery. Patients were randomly divided into three groups in radio 1:1:1 received respectively IV placebo, ibuprofen 400 mg or ibuprofen 800 mg. The first dose of study drugs was administered intravenously at the time of wound closure and then every 6 hours within 48 hours after the operation. At the end of surgical suture, 5mg morphine was injected intravenously, and then the patient-controlled intravenous analgesia pump was connected. Efficacy was assessed by morphine dosage during the first 24 hours, pain intensity score, and area under the pain-time curve after surgery. Safety was assessed by the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment was open to patients undergoing scheduled abdominal surgery (intestinal or lower abdomen) or orthopedic surgery (such as knee arthroplasty or shoulder joint reconstruction) under general anesthesia with endotracheal intubation and were expected to require patient-controlled intravenous analgesia (PCIA) pump for more than 24h for moderate to severe pain after surgery.

Exclusion Criteria:

* Those who can not understand the NRS score and cooperate with the evaluation; those who had head trauma or complicated with organic lesions of the central nervous system within 4 weeks before operation; those who developed coagulation dysfunction or took anticoagulants and antiplatelet drugs; those with a history of severe cardio-cerebrovascular disease, heart failure; those with liver and kidney dysfunction, severe endocrine system diseases, mental illness; those with a history of peptic ulcer or bleeding; those who did not control grade 2 or above hypertension or were still taking two or more of antihypertensive drugs such as angiotensin converting enzyme inhibitors (ACEI), angiotensin converting enzyme antagonists (ARB) and diuretics at admission; Increased toxicity due to the interaction of methotrexate, lithium preparations, etc. with the test drug; use of NSAIDs or analgesic muscle relaxants within 24 hours before operation, narcotic dependence or tolerance; allergy to ibuprofen or other NSAIDs; pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2020-06-10 (Estimated); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
the amount of morphine administered | during the first 24 hours
  after surgery.

SECONDARY OUTCOMES:
Pain intensity (PI) | at 0 hour,1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 18 hours, 24 hours, 30 hours, 36 hours, 42 hours and 48 hours immediately after the first administration.
  the PI was evaluated using patient self-reporting with numerical rating scales (NRS) (0= no pain to 10= intense pain)
The area under the PI-time curve (AUC) | across 3 time periods (1-24 hours, 6-24 hours, 12-24 hours)
  at rest and with movement
Total frequency and effective frequency of PCA | within 24 hours
  after surgery
Treatment failure rate | within 24 hours after the operation
  the rate of using other non-morphine drugs to remedy analgesia
Patients' evaluation of the study drug | after 48 hours of medication
  excellent=5, very good=4, good=3, general=2, bad=1

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China